CLINICAL TRIAL: NCT04614467
Title: A Double-Blind, Randomized, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of CLBS16 in Subjects With Coronary Microvascular Dysfunction and Without Obstructive Coronary Artery Disease
Brief Title: A Placebo-Controlled Trial of CLBS16 in Subjects With Coronary Microvascular Dysfunction
Acronym: FREEDOM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLBS16-P02
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Coronary Microvascular Dysfunction; Coronary Microvascular Disease; Microvascular Coronary Artery Disease
Keywords: angina; CMD; MVD; non-obstructive coronary artery disease
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GCSF-mobilized autologous CD34+ cells (Experimental)
  Interventions: Biological: CLBS16
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CLBS16 — GCSF-mobilized autologous CD34+ cells
  Arms: GCSF-mobilized autologous CD34+ cells
Biological: Placebo — isotonic solution (no CD34+ cells)
  Arms: Placebo

SUMMARY:
This clinical trial will explore the efficacy and safety of GCSF-mobilized autologous CD34+ cells for the treatment of CMD in adults currently experiencing angina and with no obstructive coronary artery disease. Eligible subjects will receive a single administration of CLBS16 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age ≥18
* History of and currently experiencing angina at least 3 times per week
* Prior diagnosis of CMD based on coronary flow reserve (CFR) ≤ 2.5 or other measures
* Canadian Cardiovascular Society (CCS) class II, III or IV chronic refractory angina
* No obstructive coronary artery disease
* On stable medical therapy for at least 30 days prior to enrollment
* Must agree to use a reliable and acceptable method of contraception for the duration of participation
* Written informed consent

Exclusion Criteria:

* Myocardial infarction within 90 days
* Prior evidence of obstructive heart disease including PCI or CABG (or planned PCI or CABG)
* Diagnosis of other specific cardiac disease
* Must meet LVEF and GFR requirements
* Current use of coumadin or DOACs
* Hypersensitivity to GCSF, apheresis or study product components
* Positive for HIV, hepatitis B or hepatitis C
* Active inflammatory or autoimmune disease, or chronic immunosuppressive state
* Drug abuse
* Pregnant or lactating
* Malignant neoplasm within 5 years
* History of Sickle Cell Disease
* Participation in another clinical study within 90 days prior to informed consent or concurrently with this study
* Previous treatment with a CD34+ cell based therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in angina frequency | Baseline to 3 and 6 months
Change from baseline in CCS angina class | Baseline to 3 and 6 months
Change from baseline in total exercise time | Baseline to 6 months
Change from baseline in health-related quality of life (HRQoL) | Baseline to 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Buck, MD, Study Director — Lisata Therapeutics, Inc.
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida - College of Medicine/ div of Cardiovascular Medicine, Gainesville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Minneapolis Heart Institute at Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - The Christ Hospital, Cincinnati, Ohio

REFERENCES:
- [Derived] Rai B, Shukla J, Henry TD, Quesada O. Angiogenic CD34 Stem Cell Therapy in Coronary Microvascular Repair-A Systematic Review. Cells. 2021 May 8;10(5):1137. doi: 10.3390/cells10051137. PMID 34066713